CLINICAL TRIAL: NCT04047082
Title: Online Videodensitometric Assessment of Aortic Regurgitation in the Cath-Lab
Acronym: OVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Amsterdam University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick W. Serruys, Professor, Imperial College London
Other Study IDs: OVAL
Record Dates: First submitted 2019-06-24; First posted 2019-08-06 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Insufficiency; Heart Valve Diseases; Regurgitation, Aortic; Paravalvular Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative aortogram (videodensitometry) — Patients that performed TAVR will have their aortogram analysed in the cath-lab by videodensitometry (quantitative aortogram)

SUMMARY:
Following the high feasibility of analyses by core laboratory with videodensitometry determined in the ASSESS-REGURGE Registry, this is an early clinical feasibility study of online videodensitometric assessment of aortograms to quantitate aortic regurgitation (AR) in the cath lab, specifically in the setting of transcatheter aortic valve replacement (TAVR)

DETAILED DESCRIPTION:
OVAL (Online Videodensitometric Assessment of Aortic Regurgitation in the Cath-Lab) is a single centre, prospective, proof-of-principle, feasibility study performed in the Academic Medical Centre (Amsterdam). One hundred consecutive patients with aortic stenosis and indication to undergo TAVR by the Institution's Heart team are being enrolled in OVAL. All final aortograms will be performed according to predetermined acquisition protocol and analysed immediately after the acquisition in the cath-lab. All aortograms will also be analysed off-line by an independent core laboratory in the Netherlands (Cardialysis, Rotterdam, The Netherlands).

The primary endpoint of the study is the feasibility of the on-line assessment of regurgitation (percentage of analysable cases). The secondary endpoint is the reproducibility of results between the on-line assessment and the off-line analysis by the independent core laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with indication to undergo TAVR by the Institution's Heart Team.

Exclusion Criteria:

* Patients that were not considered by the Institution's heart team as eligible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic aortic stenosis, requiring valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of analysis(percentage of cases considered analyzable by videodensitometry - online) | immediately
  Feasibility of analysis (percentage of cases considered analyzable by videodensitometry - online). The investigators will assess the percentage of cases that are considered by the investigators as analyzable (i.e., that the investigators are able to perform an on-line analysis of videodensitometry).
Comparison with feasibility of ASSESS-REGURGE ( to compare the percentage of analyzable cases with the percentage of the current standard found in ASSESS-REGURGE - 95.5%) | immediately
  Since ASSESS-REGURGE has the highest feasibility of analysis with quantitative aortogram, the investigators aim to compare the present feasibility (of OVAL) with the new standard from ASSESS-REGURGE. In other words, the percentage of analyzable cases in the present study will be compared with the percentage of analyzable cases found in ASSESS-REGURGE (95.5% of analyzability).

SECONDARY OUTCOMES:
Comparison of online feasibility with core lab feasibility | immediately
  The feasibility of analysis (i.e., if a cases is considered to be analyzable by videodensitometry) will be assessed on-line by the investigators and also assessed by an academic core laboratory. The result of the feasibility of analysis (percentage of analyzable cases) will be compared between the investigators assessment (on-line) and also by the core laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Study Chair — Imperial College London; Rodrigo Modolo, MD, PhD, Principal Investigator — Amsterdam University Medical Center; Robbert de Winter, MD, PhD, Principal Investigator — Amsterdam University Medical Center
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Modolo R, van Mourik M, El Bouziani A, Kawashima H, Rosseel L, Abdelghani M, Aben JP, Slots T, Sahyoun C, Baan J, Henriques JPS, Koch KT, Vis M, Soliman O, Onuma Y, Wykrzykowska J, de Winter R, Serruys PW. Online Quantitative Aortographic Assessment of Aortic Regurgitation After TAVR: Results of the OVAL Study. JACC Cardiovasc Interv. 2021 Mar 8;14(5):531-538. doi: 10.1016/j.jcin.2020.11.014. Epub 2021 Feb 10. PMID 33582086